CLINICAL TRIAL: NCT06417593
Title: Phenotypic and Genotypic Characteristics of Pseudomonas Aeruginosa Isolates in Sohag University Hospitals
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Martina Gamil Fayez, principle investigator, Sohag University
Other Study IDs: Soh-Med-24-04-016MS
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Pseudomonas Aeruginosa Infection
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group1: Pseudomonas Aeruginosa Isolates

SUMMARY:
Isolation and identification of Pseudomonas aeruginosa using basic microbiological methods, such as Gram staining, cultivation on cetrimide agar and biochemical reactions from Samples from patients with different types of health care associated infections as urinary tract infections, infected burn, ventilator associated pneumonia, blood stream infections and surgical site infections that will be obtained under complete aseptic precautions.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients with different types of health care associated infections as urinary tract infections, infected burn, ventilator associated pneumonia, blood stream infections and surgical site infections will be obtained under complete aseptic precautions.

Exclusion Criteria:

* Any infection before 48 hours of patient admission at Hospital

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples from patients with different types of health care associated infections as urinary tract infections, infected burn, ventilator associated pneumonia, blood stream infections and surgical site infections will be obtained under complete aseptic precautions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Isolation and identification of pseudomonas aeruginosa causing different nosocomial infections. | 6 months
  Isolation and identification of Pseudomonas aeruginosa using basic microbiological methods, such as Gram staining, cultivation on cetrimide agar and biochemical reactions
Identification of antibiotic susceptibility pattern of isolated strains of pseudomonas | 6 months
  Antibiotic susceptibility testing of the isolates will be performed using disc diffusion method according to clinical laboratory standards institute (CLSI) guidelines
Detection of biofilm forming isolates | 6 months
  Detection of biofilm forming isolates by tissue culture plate method.
Detection of virulence and antibiotic resistance genes of pseudomonas aeruginosa. | 6 months
  Detection of virulence and antibiotic resistance genes by conventional Polymerase Chain Reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol